CLINICAL TRIAL: NCT00694239
Title: Evaluation of the Effect of Cardiovascular Risk Assessment in Treatment Compliance in Hypertension
Brief Title: Risk Assessment and Treat Compliance in Hypertension Education Trial
Acronym: RATCHET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other); The Physicians' Services Incorporated Foundation (Other)
Responsible Party: George Dresser, University of Western Ontario
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-07-053; 13014E (Other: REB)
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Hypertension; Dyslipidemia
Keywords: hypertension; compliance
MeSH Terms: conditions — Hypertension; Dyslipidemias; Patient Compliance

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (No Intervention): Standard Care
- A (Experimental): Risk Assessment plus standard care
  Interventions: Behavioral: Knowledge of Cardiovascular Risk Assessment

INTERVENTIONS:
Behavioral: Knowledge of Cardiovascular Risk Assessment — Knowledge of Cardiovascular Risk Assessment and risk reduction at target BP, reviewed every 3-6 months.
  Arms: A

SUMMARY:
The RATCHET study assesses if patient knowledge of estimated cardiovascular risk at current and recommended target blood pressure levels improves compliance in the management of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension (new diagnosis or established diagnosis) meeting criteria for pharmacologic therapy as defined by current guidelines

Exclusion Criteria:

* Lack of written informed consent
* Previous myocardial infarction
* Previous stroke
* Congestive heart failure
* Stage 3 or greater chronic kidney disease
* Pregnancy
* Usage of medication bubble/blister package

Ages: 30 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Medication Compliance | 1 year

SECONDARY OUTCOMES:
Patient perception of cardiovascular risk | 1 year
Pilot Feasibility Study | 1 year
Blood Pressure | 1 year
Cholesterol Level | 1 year
Framingham Risk Score (stroke and coronary artery disease) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bryan J Har, MD, Principal Investigator — Western University, Canada; George K Dresser, PhD, MD, Principal Investigator — Western University, Canada
Locations (1):
- University of Western Ontario, London, Ontario, Canada

REFERENCES:
- See also: Physicians Services Incorporated — http://www.psifoundation.org/
- See also: University of Western Ontario — http://www.uwo.ca